CLINICAL TRIAL: NCT02844738
Title: Safety and Effectiveness of Autologous Regenerative Cell Therapy on Pain and Inflammation Associated With Osteoarthritis of the Shoulder
Brief Title: Safety & Effectiveness of Autologous Regenerative Cell Therapy on Pain & Inflammation of Osteoarthritis of the Shoulder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VivaTech International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ￼ IRCM-2016-113
Record Dates: First submitted 2016-07-08; First posted 2016-07-26 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- StroMed + platelet rich plasma (PRP) (Experimental): Because no enzymes or drugs are added with this mechanical process, the resulting (StroMed) cell concentrate still contains the extra-cellular matrix. In addition, the cells have not been altered by manipulation with enzymes or culturing. This autologous, cell concentrate is of minimal risk to the patient with no artificial ingredients added. Additional treatments with Platelet Rich Plasma processed by the RegenLab (RegenKit BCT-3) PRP product and by direct injection to affected joint.
  Interventions: Biological: [StroMed + platelet rich plasma (PRP)]

INTERVENTIONS:
Biological: [StroMed + platelet rich plasma (PRP)] — Patients will be treated with autologous StroMed obtained by the Adipose Ultrasonic Cell Recovery Unit and Platelet Rich Plasma processed by the RegenLab (RegenKit BCT-3) PRP product each as direct injections to the affected joints at the time of initial treatment. Thereafter the affected joints will be treated as direct injections to the joint with Platelet Rich Plasma processed by the RegenLab (RegenKit BCT-3) PRP product. Day 0 [StroMed + platelet rich plasma (PRP)], Days 7 and 14 [PRP]

SUMMARY:
This is a prospective open-label clinical study of 50 patients to determine safety and treatment potential of autologous cell therapy for pain and inflammation associated with Osteoarthritis of the shoulder. Follow-up will consist of a larger sample including 4,000 patients.

DETAILED DESCRIPTION:
This is a prospective open-label clinical study of 50 patients to determine safety and treatment potential of autologous cell therapy for pain and inflammation associated with Osteoarthritis of the shoulder. Follow-up will consist of a larger sample including 4,000 patients.

Patients will be treated for Osteoarthritis (OA) of the shoulder due to degeneration or chronic injury. They will be treated with autologous Stromed obtained by the Adipose Ultrasonic Cell Recovery Unit (AUCRU) and Platelet Rich Plasma (PRP) processed by the RegenLab (RegenKit BCT-3) PRP product each as direct injections to the affected joints. Patient outcomes will be tracked with laboratory tests for inflammation markers, the DASH and SPADI questionnaires and a follow up MRI at various endpoints to 6 months. SF-36 forms (a quality of life measure) and numerical ratings scales (NRS) will also be used to assess safety and efficacy of treatment, as well as any reduction in patient medication and/or delay in pending shoulder planning/replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with indication of Osteoarthritis. Can be from degeneration or chronic injury.
2. Patients range from 18-90 years of age.
3. Patients must be able to comply with treatment plan, laboratory tests and periodic interviews.
4. Patients with adequate renal function, Creatinine ≤ 1.5 mg/dl.
5. Patients with adequate cardiac and respiratory function.
6. Patients with adequate blood coagulation activity, PT(INR) < 1.5, APTT
7. Patients must have adequate immune system function, with no known immunodeficiency disease.
8. Greater than 6 months shoulder pain with the index side (left or right shoulder).

Exclusion Criteria:

1. Neoplastic cancer within 5 years prior to screening, except for cutaneous basal cell or squamous cell cancer resolved by excision
2. Presence of clinically significant acute or unstable cardiovascular, cerebrovascular (stroke)..
3. Diagnosis of a transient ischemic attack in the 6 months prior to screening.
4. Patients infected with hepatitis B, C or HIV.
5. Patients with Body Mass Index (BMI) > 40kg/m2
6. Presence of active infection.
7. Any other illness, psychiatric disorder, alcohol or chemical dependence that in the opinion of the investigator would render a patient unsuitable to participate in the study.
8. Conditions/therapies/factors which could confound or interfere with the evaluation of pain/mobility including, but not limited to:

   1. Treatments with strong opioid drugs in the previous 4 weeks for other pain rather than shoulder osteoarthritis
   2. Corticosteroid injection at treatment site within 1 month
   3. Consistent use of NSAIDs within 48 hours of procedure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change is being assessed for the DASH Survey (Disabilities of the Arm, Shoulder, Hand | 0,2,6 months
  Disabilities of the Arm, Shoulder, and Hand

SECONDARY OUTCOMES:
Change is being assessed by MRI of afflicted joint | 0 and (6 months optional)
  Looking for cartilage regrowth via MRI
Change is being assessed for the SPADI Survey (Shoulder Pain and Disability Index) | 0,2,6 Months
  Shoulder Pain and Disability Index
Change is being assessed for the SF36 Survey (Short Form Health Survey) | 0,2,6 Months
  Short Form Health Survey
Change is being assessed for the NRS Survey (Numerical Rating Scale for Pain) | 0,2,6 Months
  Numerical Rating Scale for Pain

CONTACTS AND LOCATIONS:
Overall Officials: Mark LoDico, MD, Principal Investigator — Advanced Regenerative Medicine
Locations (1):
- VivaTech International, Inc., Grove City, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
VivaTech will monitor data and decide if/when data can be shared

REFERENCES:
- See also: Company Website — http://www.vivatechusa.com